CLINICAL TRIAL: NCT04649905
Title: Psychological Response and Readiness to Return to Sports Associated With the Diagnosis and Treatment of Osteochondritis Dissecans of the Knee
Brief Title: Psychological Response and Readiness Associated With OCD of the Knee
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Matthew Milewski, Assistant Professor of Orthopedic Surgery, Harvard Medical School, Boston Children's Hospital
Other Study IDs: IRB-P00036878
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Osteochondritis Dissecans Knee; Psychological Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgical Treatment: Patient's in this cohort will undergo surgical treatment for OCD of the knee.
  Interventions: Procedure: Surgical Treatment
- Nonoperative Treatment: Patient's in this cohort will undergo nonoperative treatment for OCD of the knee.
  Interventions: Procedure: Nonoperative Treatment

INTERVENTIONS:
Procedure: Surgical Treatment — Surgical standard-of-care treatment for knee OCD
  Groups: Surgical Treatment
Procedure: Nonoperative Treatment — Nonoperative standard-of-care treatment for knee OCD
  Groups: Nonoperative Treatment

SUMMARY:
This study primarily aims to determine whether patients diagnosed with osteochondritis dissecans (OCD) of the knee experience psychological stress due to their diagnosis and treatment plan. Secondarily, this study aims to determine whether knee OCD patients experience a change in stress and depression as they progress through their standard-of-care treatment plan, and whether they have impaired psychological readiness for return to sport.

DETAILED DESCRIPTION:
Young athletes with poor psychological responses to injury and recovery may be at risk for suboptimal rehabilitation and return to sports. The issues of psychological readiness and fear/anxiety of reinjury are well documented in the treatment of ACL injuries in young athletes. To the investigative team's knowledge, no studies have examined the psychological response and psychological readiness to return to sports in pediatric and adolescent patients undergoing treatment for osteochondritis dissecans (OCD) of the knee.

OCD is a focal, idiopathic alteration of subchondral bone with risk for instability and disruption of adjacent articular cartilage that may result in premature osteoarthritis. It generally affects a young population between 6 and 19 years of age, with highest prevalence between the ages of 12 and 19 years of age. This condition can be treated both conservatively and surgically depending on the age of the patient, size of the lesion, severity and instability of the bone & cartilage, and previous treatment. The unclear etiology of this condition, the delayed / prolonged pre-diagnosis symptoms, varied treatment options, and unpredictable healing timelines are all factors that families and patients find frustrating about this condition. The investigators of this study believe that this leads to higher than normal psychological stress at the time of diagnosis and throughout treatment of this condition.

Improved understanding of the psychological stress and readiness to return to sport in the treatment of knee OCD can help patients, their families, and clinicians alike. Awareness can help clinicians provide the appropriate outreach and counseling for patients at risk for increased psychological stress. Improved psychological states and readiness can improve both physical and mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 11-19
* Diagnosis of knee OCD confirmed by X-ray or MRI

Exclusion Criteria:

* Had previous surgical treatment for their knee OCD lesion
* Received knee OCD non-operative treatment on the ipsilateral side for >6 months and taken out of sports/physical activities
* Guardian not comfortable with child completing survey
* Is not fluent in English

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who meet eligibility criteria presenting to either 1) Boston Children's Sports Medicine and seen by Dr. Matthew Milewski, MD, or Dr. Melissa Christino, MD, with a new diagnosis of an OCD lesion of the knee; or 2) Texas Scottish Rite Hospital's Sports Medicine Clinic and seen by Dr. Henry Ellis, MD, or Dr. Philip Wilson, MD.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
THE CHILDREN'S IMPACT OF EVENT SCALE (CRIES-13) score | Time of surgical consultation/diagnosis for knee OCD
  A CRIES-13 score is a continuous number between 0 and 65 (the higher the score, the more severe the outcome). CRIES items will be keyed to the diagnosis and treatment of OCD (i.e., the patient is asked to indicate how frequently each comment was true for them during the past 7 days with respect to their experience with OCD).
  The CRIES is a 13-item, 4-point scale assessing psychological distress. It has three subscales: intrusion, avoidance, and arousal. It is based off the Impact of Event Scale (IES) and is designed to address misinterpretation of items by children on the IES. It is designed for children 8 years of age and above to read independently. If the score is greater than or equal to 30, the score is indicative of increased subjective stress.

SECONDARY OUTCOMES:
THE CHILDREN'S IMPACT OF EVENT SCALE (CRIES-13) score | Scores taken repeatedly overtime between diagnosis and follow-up (at every clinic visit as well as 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis)
  A CRIES-13 score is a continuous number between 0 and 65 (the higher the score, the more severe the outcome). CRIES items will be keyed to the diagnosis and treatment of OCD (i.e., the patient is asked to indicate how frequently each comment was true for them during the past 7 days with respect to their experience with OCD).
  The CRIES is a 13-item, 4-point scale assessing psychological distress. It has three subscales: intrusion, avoidance, and arousal. It is based off the Impact of Event Scale (IES) and is designed to address misinterpretation of items by children on the IES. It is designed for children 8 years of age and above to read independently. If the score is greater than or equal to 30, the score is indicative of increased subjective stress.
Patient-Reported Outcomes Measurement Information System (PROMIS) Psychological Stress Experiences | Scores taken repeatedly overtime between diagnosis and follow-up (at every clinic visit as well as 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis)
  Assesses the thoughts or feelings about the world in the context of environmental or internal challenges. Patients will complete at the time of enrollment, any additional clinical visit, including 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis. There are 19 questions that are rated on a 1-5 scale. Overall, this outcome measure is scored 18-95 (lower score = less stress). Raw scores are then converted into T-scores. The investigators expect scores to increase during the early stages of treatment by at least 5 points (MCID) in the first 3 months and then decrease over time returning to baseline or above at 1- to 2-year follow up post diagnosis.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Symptoms | Scores taken repeatedly overtime between diagnosis and follow-up (at every clinic visit as well as 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis)
  This questionnaire assesses for anxiety in children and adolescents (ages 11-17). Patients will complete at the time of enrollment, any additional clinical visit, including 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis. There are 8 questions that are rated on a 1-5 scale. Overall, this outcome measure is scored 14-70 (higher score = greater severity in depression). Raw scores are then converted into T-scores. The investigators expect scores to increase during the early stages of treatment by at least 5 points (MCID) in the first 3 months and then decrease over time returning to baseline or above at 1- to 2-year follow up post diagnosis.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depressive Symptoms | Scores taken repeatedly overtime between diagnosis and follow-up (at every clinic visit as well as 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis)
  This questionnaire assesses for depression in children and adolescents (ages 11-17). Patients will complete at the time of enrollment, any additional clinical visit, including 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis. There are 8 questions that are rated on a 1-5 scale. Overall, this outcome measure is scored 14-70 (higher score = greater severity in depression). Raw scores are then converted into T-scores.
ACL-Return to Sports after Injury (ACL-RSI) | Scores taken repeatedly overtime between diagnosis and follow-up (at every clinic visit as well as 3 months, 6 months, 9 months, 1 year, and 2 years post diagnosis)
  Questionnaire used to measure the psychological impact of returning to sport after ACL reconstruction surgery. Patients will complete this questionnaire at the clinic visit when they are cleared to RTS, 1 year and 2 years post diagnosis. There are 12 questions that are rated on a 0-10 scale. Overall, this outcome measure is scored 0-100 (higher score = more psychologically ready to RTS). A score greater than or equal to 77% indicates that the patient is psychologically ready to RTS.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Milewski, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Texas Scottish Rite Hospital, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No